CLINICAL TRIAL: NCT04886479
Title: Comparing Habitual Daily Disposable Silicone Hydrogel (DDSH) Contact Lens Wearers to Habitual Daily Disposable Hydrogel (DDH) Contact Lens Wearers and Non-lens Wearers
Brief Title: Comparing Silicone Hydrogel Contact Lens Wearers to Hydrogel Contact Lens Wearers and Non-lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EX-MKTG-89
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Results first posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2023-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Daily Disposable Silicone Hydrogel Contact Lens Wearers (Experimental): Participants wore Test Lens for 3 hours
  Interventions: Device: Test Lens
- Daily Disposable Hydrogel Contact Lens Wearers (Experimental): Participants wore Test Lens for 3 hours
  Interventions: Device: Test Lens
- Non-lens Wearers (Active Comparator): Participants did not receive Test Lens
  Interventions: Other: Control

INTERVENTIONS:
Other: Control — No lens
  Arms: Non-lens Wearers
Device: Test Lens — Low Dk HEMA contact lens worn for 3 hours
  Arms: Daily Disposable Hydrogel Contact Lens Wearers; Daily Disposable Silicone Hydrogel Contact Lens Wearers

SUMMARY:
This study was a multi-site, prospective, randomized, non-masked, unilateral, non-dispensing study.

DETAILED DESCRIPTION:
The purpose of this study was to to compare physiological response baseline data between 3 groups - habitual wearers of Daily Disposable Silicone Hydrogel (DDSH) contact lenses, habitual wearers of Daily Disposable Hydrogel (DDH) contact lenses, and non-lens wearers. The study then compared physiological response data following wear of a low Dk HEMA contact lens between habitual wearers of DDSH and habitual wearers of DDH.

ELIGIBILITY:
Inclusion Criteria:

1. Is between 17 and 60 years of age inclusive (age matching required between all 3 study groups), and has full legal capacity to volunteer;
2. Has had a self-reported oculo-visual examination in the last two years.
3. Has read and signed an information consent letter;
4. Is willing and able to follow instructions and maintain the appointment schedule;
5. No previous history of overnight contact lens wear or PMMA (polymethylmethacrylate) lens wear.
6. Auto-refraction vertexed spherical equivalent between +4.00 and -8.00 (prescription matching required between groups 1 & 2). This criterion is non-applicable to participants in group 3.
7. Is found to be in one of the study groups matched by age (±5 years), ethnicity (Asian vs. non-Asian) and CL Rx (±2.00 D) according using the following criteria.

   GROUP 1: For the past (minimum) 6 months has ONLY worn spherical DDSH lenses AND prior to wearing this lens they only wore SH material lenses in the past (minimum) 3 total years.

   GROUP 2: For the past (minimum) 6 months has ONLY worn spherical DDH lenses AND prior to wearing this lens they only wore H material lenses in the past (minimum) 3 total years.
8. For groups 1 & 2, currently and for at least the previous 6 months has had habitual daily disposable wear schedule of at least 8 hrs a day, 5 days a week in only one material category - either silicone hydrogel or hydrogel material. This criterion is not-applicable to participants in group 3.
9. Is willing to wear the study contact lens in the randomized eye for 3 hours of eye closure on the second study day. This criterion is not-applicable to participants in group 3.
10. Has clear and healthy corneas and anterior eye and no active ocular disease;
11. Can achieve monocular HCVA of logMAR 0.10 or better in each eye with subjective refraction or pinhole.
12. Can achieve acceptable fit and comfort in the randomized eye with the study lens. This criterion will be confirmed at the baseline visit (V1). This criterion is not-applicable to participants in group 3.
13. Has a wearable pair of spectacles.

Exclusion Criteria:

1. Is participating in any concurrent clinical trial;
2. Is unable/unwilling to provide permission for the study site to seek CL history from their eye care practitioner
3. Has any known active ocular disease and/or infection;
4. Has a systemic condition that in the opinion of the investigator may affect a study measure or interfere with contact lens wear; this may include, but not be limited to, diabetes, hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes, and systemic connective tissue disorders e.g. rheumatoid arthritis.
5. Is using any systemic or topical medications that in the opinion of the investigator may affect a study measure;
6. Has known sensitivity to fluorescein dye, topical anesthetic, or products to be used in the study;
7. Appears to have any active ocular pathology, ocular anomaly or severe insufficiency of lacrimal secretion (severe dry eye) that would affect the wearing of contact lenses;
8. Appears to have any signs of corneal inflammation or previous infection or corneal opacity/scar;
9. Is pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit), due to potential ocular physiological changes, such as changes in the corneal shape and cell types;
10. Is aphakic;
11. Has undergone refractive error surgery, or has a history of any ocular surgery or injury.
12. Is a toric or multifocal contact lens wearer.

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (2):
- CORE, University of Waterloo, Waterloo, Canada
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-six participants were screened, with 3 of these not meeting all eligibility criteria and were considered screen failures. One participant withdrew for reasons unrelated to the study. These participants were not included in the total number of participants enrolled.
Units Other Than Participants: Eyes [single]
Groups:
- DDSH Lens Wearers: Participants wore habitual DDSH Lens in both eyes for 6-8 hours (Period 1, observational). Afterwards, participants wore the Test Lens in one randomized eye that was kept closed and patched for 3 hours (Period 2, interventional).
- DDH Lens Wearers: Participants wore habitual DDH Lens in both eyes for 6-8 hours (Period 1, observational). Afterwards, participants wore the Test Lens in one randomized eye that was kept closed and patched for 3 hours (Period 2, interventional).
- Non-lens Wearers: Participants had no previous history of contact lens wear. Participants wore habitual spectacles, if any, for 6-8 hours (Period 1, observational). They did not receive the Test Lens and were not involved in Period 2.
Period: Period 1: Habitual Device, 6-8 Hours
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers
Started | 10; 20 Eyes [single] | 3; 6 Eyes [single] | 9; 18 Eyes [single]
Completed | 10; 20 Eyes [single] | 3; 6 Eyes [single] | 9; 18 Eyes [single]
Not Completed | 0; 0 Eyes [single] | 0; 0 Eyes [single] | 0; 0 Eyes [single]
Period: Period 2: Test Lens, 3 Hours
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers
Started | 10; 10 Eyes [single] | 3; 3 Eyes [single] | 0; 0 Eyes [single] (None of the participants in the control group were involved in Period 2)
Completed | 10; 10 Eyes [single] | 3; 3 Eyes [single] | 0; 0 Eyes [single]
Not Completed | 0; 0 Eyes [single] | 0; 0 Eyes [single] | 0; 0 Eyes [single]

BASELINE CHARACTERISTICS:
Groups:
- DDSH Lens Wearers: Participants who habitually wear DDSH lenses
- DDH Lens Wearers: Participants who habitually wear DDH lenses
- Non-lens Wearers: Participants that do not wear either DDSH or DDH Lens.
- Total: Total of all reporting groups
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers | Total
Number analyzed (Participants) | 10 | 3 | 9 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (13.2) | 30.0 (7.5) | 31.7 (13.2) | 31.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 6 | 13
  Male | 5 | 1 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity was measured due to possible differences in physiological response to corneal hypoxia in Asian and non-Asian participants. All subjects in this study were of non-Asian ethnicity, due to difficulty in finding and recruiting Asian candidates at the study site.
  Participants
    Non-Asian | 10 | 3 | 9 | 22
    Asian | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Limbal Redness - DDSH, DDH, Non-lens Groups
Description: Objective grading (0-4, severity increases in 0.1 steps; 0=no redness, 4=severe redness) of limbal redness after 6-8 hours of habitual device wear. For each participant, measurements were taken for both eyes (OD - right eye, OS - left eye) at two locations (T - temporal, N - nasal).
Time Frame: 6-8 hours of habitual wear
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes (single)
Groups:
- DDSH Lens Wearers: Participants wore habitual DDSH Lens in both eyes
- DDH Lens Wearers: Participants wore habitual DDH Lens in both eyes
- Non-lens Wearers: Participants did not wear either DDSH or DDH Lens
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers
Number analyzed (Participants) | 10 | 3 | 9
Number analyzed (Eyes (single)) | 20 | 6 | 18
score on a scale
  OD, T | 0.41 [0.24 to 0.58] | 0.37 [0.05 to 0.68] | 0.44 [0.26 to 0.63]
  OD, N | 0.49 [0.25 to 0.73] | 0.40 [-0.04 to 0.84] | 0.44 [0.19 to 0.70]
  OS, T | 0.54 [0.35 to 0.73] | 0.30 [-0.05 to 0.65] | 0.46 [0.25 to 0.66]
  OS, N | 0.32 [0.18 to 0.46] | 0.37 [0.12 to 0.62] | 0.41 [0.27 to 0.56]

2. Primary Outcome: Bulbar Redness DDSH, DDH, Non-lens Groups
Description: Objective grading (0-4, severity increases in 0.1 steps; 0=no redness, 4=severe redness) of bulbar redness after 6-8 hours of habitual device wear. For each participant, measurements were taken for both eyes (OD - right eye, OS - left eye) at two locations (T - temporal, N - nasal).
Time Frame: 6-8 hours of habitual wear
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes (single)
Groups:
- Non-lens Wearers: Participants did not wear DDSH or DDH Lens
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers
Number analyzed (Participants) | 10 | 3 | 9
Number analyzed (Eyes (single)) | 20 | 6 | 18
score on a scale
  OD, T | 0.76 [0.55 to 0.97] | 0.67 [0.28 to 1.05] | 0.79 [0.56 to 1.01]
  OD, N | 0.86 [0.59 to 1.13] | 0.83 [0.33 to 1.33] | 0.71 [0.42 to 1.00]
  OS, T | 0.93 [0.63 to 1.23] | 0.73 [0.18 to 1.28] | 0.80 [0.48 to 1.12]
  OS, N | 0.86 [0.60 to 1.12] | 0.60 [0.13 to 1.07] | 0.67 [0.40 to 0.94]

3. Primary Outcome: Limbal Vessel Ingrowth - DDSH, DDH, Non-lens Groups
Description: Number of participants with limbal vessel ingrowth longer than 0.50 mm at any of the 4 corneal quadrants (superior, inferior, nasal, temporal) after 6-8 hours of device wear.
Time Frame: 6-8 hours of habitual wear
Measure: Count of Participants; unit: Participants
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers
Number analyzed (Participants) | 10 | 3 | 9
Participants | 2 | 2 | 0

4. Primary Outcome: Limbal Redness - DDSH, DDH Groups
Description: Objective grading (0-4, severity increases in 0.1 steps; 0=no redness, 4=severe redness) of limbal redness by location (T - temporal, N - nasal) and time (t). Measurements were taken at baseline and over a 3 hour period of closed-eye Test Lens wear.
Time Frame: Immediately upon eye opening (t=baseline) and lens removal (t=0), 1 hour (t=1), and 3 hours (t=3) post lens removal
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes (single)
Groups:
- DDSH Lens Wearers: Habitual DDSH lens wearers wore the Test Lens in one randomized eye that was kept closed and patched for 3 hours. The contralateral eye remained open.
- DDH Lens Wearers: Habitual DDH lens wearers wore the Test Lens in one randomized eye that was kept closed and patched for 3 hours. The contralateral eye remained open.
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers
Number analyzed (Participants) | 10 | 3
Number analyzed (Eyes (single)) | 10 | 3
score on a scale
  T, t=baseline | 0.48 [0.28 to 0.68] | 0.33 [-0.04 to 0.71]
  T, t=0 hour | 0.70 [0.50 to 0.90] | 0.43 [0.07 to 0.79]
  T, t=1 hours | 0.61 [0.36 to 0.86] | 0.43 [-0.03 to 0.90]
  T, t=3 hours | 0.71 [0.45 to 0.97] | 0.30 [-0.17 to 0.77]
  N, t=baseline | 0.36 [0.16 to 0.56] | 0.50 [0.13 to 0.87]
  N, t=0 hour | 0.72 [0.44 to 1.00] | 0.63 [0.11 to 1.15]
  N, t=1 hours | 0.57 [0.33 to 0.81] | 0.57 [0.13 to 1.01]
  N, t=3 hours | 0.63 [0.34 to 0.92] | 0.43 [-0.10 to 0.97]

5. Primary Outcome: Bulbar Redness - DDSH, DDH Groups
Description: Objective grading (0-4, severity increases in 0.1 steps; 0=no redness, 4=severe redness) of bulbar redness by location (T - temporal, N - nasal) and time (t). Measurements were taken at baseline and over a 3 hour period of closed-eye Test Lens wear.
Time Frame: Immediately upon eye opening (baseline) and lens removal (t=0), 1 hour (t=1), and 3 hours (t=3) post lens removal
Measure: Mean (95% Confidence Interval); unit: score on a scale
Units Other Than Participants: Eyes (single)
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers
Number analyzed (Participants) | 10 | 3
Number analyzed (Eyes (single)) | 10 | 3
score on a scale
  T, t=baseline | 0.87 [0.55 to 1.19] | 0.60 [0.02 to 1.18]
  T, t=0 hour | 1.00 [0.73 to 1.27] | 0.63 [0.14 to 1.12]
  T, t=1 hours | 0.89 [0.51 to 1.27] | 0.57 [-0.12 to 1.25]
  T, t=3 hours | 1.03 [0.69 to 1.37] | 0.60 [-0.03 to 1.23]
  N, t=baseline | 0.78 [0.47 to 1.09] | 0.80 [0.23 to 1.37]
  N, t=0 hour | 1.14 [0.87 to 1.41] | 0.87 [0.37 to 1.36]
  N, t=1 hours | 1.00 [0.73 to 1.27] | 0.73 [0.24 to 1.23]
  N, t=3 hours | 1.21 [0.81 to 1.61] | 0.77 [0.03 to 1.50]

6. Secondary Outcome: Central Corneal Swelling (%) - DDSH, DDH Groups
Description: Difference in central corneal swelling (μm, Visante OCT) at baseline (before lens insertion) vs. measurements taken over a 3 hour period following Test Lens removal. Derived by the formula: corneal swelling % = (measured corneal thickness - baseline corneal thickness) x 100 /baseline corneal thickness.
Time Frame: Immediately upon eye opening and lens removal (t=0), 0.5 hours (t=0.5), 1 hour (t=1), 2 hours (t=2), and 3 hours (t=3) post lens removal
Measure: Mean (95% Confidence Interval); unit: Percent change in corneal swelling (%)
Units Other Than Participants: Eyes (single)
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers
Number analyzed (Participants) | 10 | 3
Number analyzed (Eyes (single)) | 10 | 3
Percent change in corneal swelling (%)
  t=0 hours | 9.67 [7.28 to 12.07] | 9.34 [4.97 to 13.71]
  t=0.5 hours | 7.68 [5.61 to 9.75] | 6.82 [3.03 to 10.60]
  t=1 hour | 5.17 [3.57 to 6.76] | 4.26 [1.35 to 7.17]
  t=2 hours | 0.98 [0.20 to 1.77] | 0.45 [-0.99 to 1.88]
  t=3 hours | -0.41 [-1.15 to 0.32] | -0.45 [-1.80 to 0.89]

ADVERSE EVENTS:
Time Frame: Through study exit, up to 30 days from the first visit.
Groups:
- DDSH Lens Wearers: Participants that wore DDSH Lens in Period 1 and Test Lens in Period 2
- DDH Lens Wearers: Participants that wore DDH Lens in Period 1 and Test Lens in Period 2
- Non-lens Wearers: Participants that did not wear DDSH or DDH Lenses in Period 1
Arm/Group | DDSH Lens Wearers | DDH Lens Wearers | Non-lens Wearers
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/3 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DDSH Lens Wearers (N=10) | DDH Lens Wearers (N=3) | Non-lens Wearers (N=9)
Lightheadedness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — Transitional feeling of light-headedness during confocal microscopy. Unrelated to study, as neither DDH Lens nor DDSH Lens were worn at time of event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04886479/Prot_SAP_000.pdf